CLINICAL TRIAL: NCT00266240
Title: A Randomized, Double-blind Study to Determine the Effect of GK Activator (2) on Efficacy (HbA1c), Safety, Tolerability and Pharmacokinetics in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of GK Activator (2) in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM18248
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: GK Activator (2)
- 2 (Experimental)
  Interventions: Drug: GK Activator (2)
- 3 (Experimental)
  Interventions: Drug: GK Activator (2)
- 4 (Experimental)
  Interventions: Drug: GK Activator (2)
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GK Activator (2) — Escalating doses po bid
  Arms: 1; 2; 3; 4
Drug: Placebo — po bid
  Arms: 5

SUMMARY:
This study will evaluate the efficacy, safety, tolerability, and pharmacokinetics of oral GK Activator (2), compared to placebo, in patients with type 2 diabetes mellitus. The anticipated time on study treatment is less than 3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 30-75 years of age;
* type 2 diabetes mellitus for >3 months before screening;
* treatment-naive, inadequately controlled diabetes despite diet and exercise, or inadequately controlled diabetes in patients on monotherapy or combination therapy (maximum of 2 oral anti-hyperglycemic medications).

Exclusion Criteria:

* type 1 diabetes mellitus;
* women who are pregnant, breast-feeding or not using adequate contraceptive methods.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2005-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
HbA1c mean change from baseline, compared to placebo. | Week 12

SECONDARY OUTCOMES:
Additional parameters of glycemic and lipid control. | Week 12
AEs, laboratory parameters. | Throughout study
Pharmacokinetic and exposure-response relationship | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- United States (19):
  - Tucson, Arizona
  - Pine Bluff, Arkansas
  - Chula Vista, California
  - Spring Valley, California
  - West Hills, California
  - Hollywood, Florida
  - Atlanta, Georgia
  - Binghamton, New York
  - Fayetteville, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Springdale, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Beaver, Pennsylvania
  - Tipton, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Plano, Texas
  - Renton, Washington
- Bulgaria (4):
  - Dimitrovgrad
  - Pleven
  - Rousse
  - Sofia
- Zagreb, Croatia
- Guatemala City, Guatemala
- Hungary (3):
  - Budapest
  - Győr
  - Kecskemét
- Mexico (4):
  - Chihuahua City
  - Cuernavaca
  - Durango
  - Mexico City
- Poland (5):
  - Bialystok
  - Gdansk
  - Gorzów
  - Krakow
  - Wroclaw